CLINICAL TRIAL: NCT03557502
Title: Heat Therapy Versus Exercise Training in Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UOregon
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2022-09

CONDITIONS: Hypertension; Cardiovascular Diseases; Arterial Hypertension
Keywords: Stage 1 hypertension; Arterial Stiffness
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized parallel study design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat Therapy Group (Experimental): Group will undergo 30 sessions of heat therapy over approximately 10 weeks. Sessions will require subjects to be immersed in hot water for up to 45 minutes per session.
  Interventions: Other: Heat Therapy Group
- Aerobic Exercise Group (Experimental): Group will undergo 30 sessions of aerobic exercise training over approximately 10 weeks. Sessions will require subjects to exercise on a cycle ergometer for up to 45 minutes per session.
  Interventions: Other: Aerobic Exercise Group

INTERVENTIONS:
Other: Heat Therapy Group — 30 sessions of immersion in 40.5 degree celsius water for 45 minutes per session
  Arms: Heat Therapy Group
Other: Aerobic Exercise Group — 30 sessions of aerobic exercise training for 45 minutes at 60% of VO2peak
  Arms: Aerobic Exercise Group

SUMMARY:
This is a clinical trial to determine whether 30 sessions of heat therapy in the form of hot water immersion is better than 30 sessions of traditional aerobic exercise training on blood pressure reduction in people with elevated or Stage 1 hypertension.

DETAILED DESCRIPTION:
Hypertension accounts for more cardiovascular disease related deaths than any other modifiable risk factor. While exercise training can be effective at reducing blood pressure in some individuals, many people do not respond to exercise training, and many more are unwilling to undergo regular exercise training. Alternative options need to be explored. This is a clinical trial to determine whether 30 sessions of heat therapy in the form of hot water immersion is better than 30 sessions of traditional aerobic exercise training on blood pressure reduction in people with elevated blood pressure (hypertension). The investigators will evaluate known biomarkers of cardiovascular health. It is hypothesized that heat therapy will be superior to exercise training on blood pressure reduction.

ELIGIBILITY:
Inclusion Criteria:

* Systolic Blood Pressure 120 mmHg or greater and less than 180 mmHg or Diastolic Blood Pressure of 80mmHg or greater and less than 120mmHg

Exclusion Criteria:

* Secondary hypertension; diagnosed cardiovascular disease other than hypertension; taking anti-hypertensive drugs; BMI of 35 or greater; fasting glucose greater than 125 mg/dl; women who are pregnant, nursing, or desiring to become pregnant.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T Minson, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be placed in Research Electronic Data Capture (REDCap)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year following completion of subject testing
Access Criteria: Access to REDCap
URL: http://www.project-redcap.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three enrollees declined to participate after being registered for the clinical trial (assigned a participant number) but before initiating the intervention.
Pre-assignment Details: Protocol 2 participants consisted of a subset of participants from Protocol 1 (i.e. Participants were only eligible for Protocol 2 if they participated in Protocol 1). Not all participants who participated in Protocol 1 were qualified or interested to participate in Protocol 2.
Period: Protocol 1
Arm/Group | Heat Therapy Group | Aerobic Exercise Group
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0
Period: Protocol 2
Arm/Group | Heat Therapy Group | Aerobic Exercise Group
Started | 17 | 14
Completed | 15 | 12
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Met exclusion criteria at Post timepoint | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Aerobic Exercise Group: Group will undergo 30 sessions of aerobic exercise training over approximately 10 weeks. Sessions will require subjects to exercise on a cycle ergometer for up to 45 minutes per session.
  Aerobic Exercise Group: 30 sessions of aerobic exercise training consisting of a 5-minute warm-up of seated upright cycling at 30% VO2 peak, followed by 40 minutes of cycling at 60% VO2 peak, then a 5-minute cool down at 30% VO2 peak.
- Total: Total of all reporting groups
Arm/Group | Heat Therapy Group | Aerobic Exercise Group | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 47.57 [36 to 59] | 47.95 [35 to 60] | 47.76 [35 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 19 | 17 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Reduction: Change in Systolic and Diastolic Ambulatory Blood Pressure (mmHg) After 30 Sessions of Intervention
Description: Ambulatory blood pressure (ABP) was measured at baseline (PRE) and after 30 heat therapy or exercise training sessions (POST) over the course of 8-10 weeks. Two individuals performed post-intervention testing after completing only 27 sessions (1 in each group). Participants arrived at the lab and were fitted with an oscillometric blood pressure cuff attached to an ambulatory blood pressure monitor. The monitor was programmed to inflate and assess blood pressure every 20 min during self-reported waking hours and every 60 min during self-reported sleeping hours. Waking and sleeping times and measurement frequency were replicated at POST within each participant. Ambulatory blood pressure data were analyzed as 24-h total for both systolic and diastolic blood pressure. Change was calculated as the value at the POST timepoint minus the value at the PRE timepoint.
Time Frame: 10 weeks
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Heat Therapy Group | Aerobic Exercise Group
Number analyzed (Participants) | 21 | 20
mmHg
  Change in systolic Ambulatory Blood Pressure | -1 [-4 to 3] | 0 [-3 to 4]
  Change in diastolic Ambulatory Blood Pressure | 0 [-3 to 2] | 1 [-2 to 3]

2. Secondary Outcome: Arterial Stiffness: Change in Carotid-femoral Pulse Wave Velocity (m/s) From Pre (Baseline) to Post (After 30 Sessions of Intervention)
Description: Carotid-femoral pulse wave velocity (m/s) was measured as a marker of arterial stiffness using a pressure transducing tonometer over the carotid artery and an inflated leg cuff to detect the femoral artery pulse waveform using air displacement at baseline (PRE) and after 30 heat therapy or exercise training sessions (POST) over the course of 8-10 weeks. Two individuals performed post-intervention testing after completing only 27 sessions (1 in each group). Change was calculated as the value at the POST timepoint minus the value at the PRE timepoint.
Time Frame: 10 weeks
Measure: Mean (95% Confidence Interval); unit: meters/second
Arm/Group | Heat Therapy Group | Aerobic Exercise Group
Number analyzed (Participants) | 21 | 20
meters/second | -0.0 [-0.3 to 0.3] | -0.1 [-0.4 to 0.2]

ADVERSE EVENTS:
Time Frame: The average intervention duration for both aerobic exercise and heat therapy was 10 weeks, although the range was 8-13 weeks and 8-16 weeks, respectively.
Arm/Group | Heat Therapy Group | Aerobic Exercise Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT03557502/Prot_001.pdf
  • Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT03557502/SAP_002.pdf
  • Informed Consent Form (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT03557502/ICF_000.pdf